CLINICAL TRIAL: NCT03293160
Title: An Evaluation of the Michigan State Innovation Model in Washtenaw and Livingston Counties
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Center for Healthcare Research and Transformation (Unknown); Community Foundation of Southeast Michigan (Unknown)
Responsible Party: Principal Investigator, Brady Post, Graduate Student Research Assistant, University of Michigan
Other Study IDs: HUM00133309
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: High Utilization of Emergency Departments

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: The set of patients in the sample who are offered enrollment in care management services.
  Interventions: Other: Care management services
- Control group: The set of patients in the sample who are not initially offered enrollment in care management services (will be offered enrollment after six months).

INTERVENTIONS:
Other: Care management services — Patients who receive care management services will interact with a care manager who will take an inventory of the patient's needs (including social determinants of health such as housing) and provide guidance about available social supports and clinical resources.
  Groups: Treatment group

SUMMARY:
This study will examine the effects of a care management program on the health and health spending outcomes of patients residing in Michigan's Washtenaw and Livingston Counties.

DETAILED DESCRIPTION:
In 2017, the State of Michigan will offer enrollment in care management services to a set of patients in Washtenaw and Livingston Counties who are predicted to be high-frequency users of emergency departments. This is a quality improvement initiative. The Center for Healthcare Research and Transformation (CHRT) will administer this enrollment and collect patient data. The Principal Investigators will conduct a study that uses the data from this quality improvement initiative to compare the outcomes of the treatment and control groups. Specifically, the study will examine whether the care management services had an effect on the number of emergency department visits and the total healthcare spending of the patients in the treatment group.

The present study therefore is the second of two related projects - the first is the CHRT-administered random assignment and enrollment of patients into care management services. The present study is a secondary analysis of the data produced by the first project.

This Protocol Registration and Results submission refers to the secondary analysis component wherever applicable, and where not applicable, describes the information relevant to the CHRT project. For example, while the present study does not assign anyone into treatment or control groups, the Sample Description indicates "Probability Sample" to describe the way in which CHRT intends to enroll patients.

ELIGIBILITY:
Inclusion criteria:

1. reside in Washtenaw or Livingston counties or have an unknown address;
2. Have a probability of being admitted to an emergency department (ED) in Washtenaw or Livingston counties that exceeds a threshold value in a predictive model;

Exclusion criteria

1. Patients referred by a community provider
2. Patient declines to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who frequently use the emergency department of hospitals located in Washtenaw or Livingston Counties.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Emergency department utilization | 6 months
  Number of emergency department visits per patient

SECONDARY OUTCOMES:
Health care spending | 6 months
  Dollars of health care spending incurred by patient

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Udow-Phillips, MHSA, Study Director — Center for Healthcare Research & Transformation
Locations (1):
- Center for Healthcare Research & Transformation, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Post B, Lapedis J, Singh K, Valenstein P, Buyuktur AG, Teske K, Ryan AM. Predictive Model-Driven Hotspotting to Decrease Emergency Department Visits: a Randomized Controlled Trial. J Gen Intern Med. 2021 Sep;36(9):2563-2570. doi: 10.1007/s11606-021-06664-1. Epub 2021 Mar 10. PMID 33694072